CLINICAL TRIAL: NCT01098864
Title: Transcranial Magnetic Stimulation of the Prefrontal Cortex: Effects on Risky Decision Making and Temporal Discounting.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was withdrawn prior to the first subject being enrolled due to the Co-Investigator leaving the university
Sponsor: University of Arkansas (Other)
Responsible Party: Mark Mennemeier, PhD / Principal Investigator, UAMS
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 109639
Record Dates: First submitted 2010-01-19; First posted 2010-04-05 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Decision Making
Keywords: Behavior; Impulsivity; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Behavior; Impulsive Behavior | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: transcranial magnetic stimulation — low frequency (1 Hz) repeated transcranial magnetic stimulation will be delivered to the dorsal lateral prefrontal cortex (DLPFC) area for a period of 15 minutes to test for effect on executive function (e.g., decision choice and subjective value). Four sessions will be conducted per subject; 2 active stimulations,(1 left DLPFC, 1 right DLPFC) and 2 sham stimulations (1 left DLPFC, 1 right DLPFC) with a minimum of 48 hours between every stimulation. Pre and post stimulations measures of cognitive and executive function will be collected and analyzed for significant differences.
  Other Names: Magstim Super Rapid 2 Stimulator w/ 70mm figure eight stimulating coil

SUMMARY:
The main objective of this study is to examine the effects of magnetic stimulation on the prefrontal cortex. We plan to use low frequency, repeated transcranial magnetic stimulation (1 Hz rTMS) to temporarily inhibit activity in the prefrontal cortex and measure the resulting effect on two decision-making tasks. The prefrontal cortex is thought to mediate or control cognitive functions like decision-making, planning, memory, and inhibit impulsive behavior.Previous research has indicated that rTMS over the right dorsal lateral prefrontal cortex will lead to preferences for riskier alternatives. Our hypothesis is that rTMS over the right DLPFC will lead to greater preference for the riskier alternative and greater temporal discounting.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants willing to give informed consent to participate
* complete the Transcranial magnetic stimulation Adult Safety Screen
* have a MRI scan
* wear ear plugs during rTMS
* receive rTMS over the designated course of days
* complete cognitive assessments and decision making tasks.
* return for post-testing on all tasks after completing all rTMS sessions

Exclusion Criteria:

* Diagnosed neurological and/or psychiatric disorders requiring hospitalization or medication
* pregnancy or the possibility of pregnancy at the time of consent
* a history of tinnitus
* metal implants in head or neck or a pacemaker
* poorly-controlled migraines
* a history of head injury, stroke, previous brain neurosurgery, or loss of consciousness due to head injury lasting greater than 10 minutes
* a personal or family history of epilepsy or seizures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
The k metric of a hyperbolic function for delayed discounting | 12-18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Mennemeier, PhD, Principal Investigator — Universtiy of Arkansas for Medical Sciences